CLINICAL TRIAL: NCT05545319
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 2, DOUBLE-BLIND, 2-ARM STUDY TO INVESTIGATE ORALLY ADMINISTERED NIRMATRELVIR/RITONAVIR COMPARED WITH PLACEBO/RITONAVIR FOR THE TREATMENT OF SEVERE COVID-19 IN HOSPITALIZED PARTICIPANTS WHO ARE IMMUNOCOMPROMISED OR AT INCREASED RISK FOR SEVERE COVID-19 OUTCOMES
Brief Title: A Study to Learn About the Medicine Called Nirmatrelvir Used in Combination With Ritonavir in People With Weakened Immune Systems or at Increased Risk for Poor Outcomes Who Are Hospitalized Due to Severe COVID-19
Acronym: EPIC-HOS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination due to challenges related to the operational feasibility of the study, taking into account the current epidemiology and declining hospitalization rates for severe COVID-19.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4671031; 2022-002447-22 (EudraCT Number)
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); Coronavirus Disease 2019 (COVID-19); Immunocompromised; Hospitalization; Child, Hospitalized
Keywords: COVID-19; Respiratory Tract Infections; Infections; Pneumonia, Viral; Pneumonia; Virus Diseases; Coronavirus Infections; Coronaviridae Infections; Nidovirales Infections; Ribonucleic acid (RNA) virus Infections; Lung Diseases; Respiratory Tract Diseases; Ritonavir; HIV Protease Inhibitors; Viral Protease Inhibitors; Protease Inhibitors; Enzyme Inhibitors; Molecular Mechanisms; Pharmacological Action; Anti-human immunodeficiency virus (HIV) Agents; Anti-Retroviral Agents; Antiviral Agents; Anti-Infective Agents; Cytochrome P-450 CYP3A Inhibitors; Cytochrome P-450 Enzyme Inhibitors; Paxlovid; Nirmatrelvir
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections; Infections; Pneumonia, Viral; Pneumonia; Virus Diseases; Coronavirus Infections; Coronaviridae Infections; Nidovirales Infections; Lung Diseases; Respiratory Tract Diseases | interventions — nirmatrelvir; nirmatrelvir and ritonavir drug combination; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nirmatrelvir/ritonavir (Experimental): Participants will receive nirmatrelvir/ ritonavir 300 mg/100 mg (or 150 mg/100 mg for participants with estimated glomerular filtration rate (eGFR) or estimated creatinine clearance (eCrCl) ≥30 to <60 mL/min) every 12 hours from Day 1 through Day 15
  Interventions: Drug: Nirmatrelvir; Drug: Ritonavir
- Placebo/ritonavir (Experimental): Participants will receive placebo 0 mg/ritonavir 100 mg every 12 hours for 15 days.
  Interventions: Drug: Ritonavir; Drug: Placebo for nirmatrelvir

INTERVENTIONS:
Drug: Nirmatrelvir — Participants will receive 2 tablets of nirmatrelvir (or 1 tablet for participants with eGFR or eCrCl ≥30 to <60 mL/min) every 12 hours
  Other Names: Paxlovid
  Arms: Nirmatrelvir/ritonavir
Drug: Ritonavir — Participants will receive 1 capsule of ritonavir every 12 hours
  Other Names: Norvir
Drug: Placebo for nirmatrelvir — Participants will receive 2 tablets of placebo for nirmatrelvir (or 1 tablet for participants with eGFR or eCrCl ≥30 to <60 mL/min) every 12 hours. A placebo does not have any medicine in it but looks just like the medicine being studied.
  Arms: Placebo/ritonavir

SUMMARY:
A Study to Learn About the Medicine Called Nirmatrelvir Used in Combination With Ritonavir in People with Weakened Immune Systems or at Increased Risk for Poor Outcomes who are Hospitalized Due to Severe COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Meeting 1 of the 2 categories of COVID-19 risk:
* Category A: Immunocompromised
* Category B: Non-Immunocompromised, but with ≥2 risk factors
* Onset of signs/symptoms attributable to COVID-19 ≤10 days prior to the day of randomization for non-immunocompromised participants (Category B).
* Confirmed SARS-CoV-2 infection as determined by Reverse transcription polymerase chain reaction (RT-PCR) or acceptable test method performed by a health care provider in any specimen collected within 48 hours prior to randomization.
* Hospitalized for inpatient care for the treatment of clinical manifestations of severe COVID-19.
* Requirement for oxygen supplementation (via nasal cannula, mask, non-invasive ventilation [NIV] or high flow oxygen) to maintain SpO2 ≥94% at the time of Screening and Randomization.

Exclusion Criteria:

* Critical illness, defined by ≥1 of the following:
* Requirement for mechanical ventilation or extracorporeal membrane oxygenation (ECMO) at randomization, or likely to require intermittent mandatory ventilation (IMV) or ECMO within 12 hours of randomization .
* Multi-organ dysfunction/failure.
* Hemodynamically unstable, eg. septic shock, cardiac failure or requiring vasopressors.
* Participant not expected to survive 24 hours from time of randomization.
* History of severe chronic liver disease
* Receiving dialysis of any kind or severe renal impairment
* Use of nirmatrelvir/ritonavir as an outpatient to treat the current COVID-19 related illness ≤7 days of randomization

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-13 (Estimated); Primary Completion 2023-09-21 (Estimated); Study Completion 2024-01-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in SARS-CoV-2 RNA level in nasopharyngeal (NP) swabs | Day 1 through Day 5
  Evaluate effect of nirmatrelvir/ritonavir compared to placebo/ritonavir on SARS-CoV-2 viral RNA levels in NP swabs in hospitalized participants.

SECONDARY OUTCOMES:
Time to sustained clinical recovery. | Day 1 through Day 30
  Evaluate effect of nirmatrelvir/ritonavir compared to placebo/ritonavir treatment on clinical outcomes when added to background usual care, for the treatment of severe COVID-19 in hospitalized participants.
  Time to sustained clinical recovery is defined as the first day during the 30 days after randomization in which a participant attains a score of 1, 2, or 3 on the 8-point ordinal scale (ie, remains alive and is either not hospitalized or is hospitalized but no longer requires ongoing inpatient medical care for COVID-19) for at least 7 consecutive days.
Proportion of participants with death from any cause or initiation of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | Day 1 through Day 30
  Evaluate effect of nirmatrelvir/ritonavir compared to placebo/ritonavir treatment on clinical outcomes when added to background usual care, for the treatment of severe COVID-19 in hospitalized participants.
Proportion of participants with SARS-CoV-2 RNA <Lower Limit of Quantitation (<LLOQ) (defined as <2.0 log10 copies/mL) in NP swabs | Day 1 through Day 15
  Evaluate effect of nirmatrelvir/ritonavir compared to placebo/ritonavir on SARS-CoV-2 viral RNA levels in NP swabs in hospitalized participants.
Proportion of participants with sustained NP swab SARS-CoV-2 RNA <LLOQ (defined as <2.0 log10 copies/mL) | Day 15 through Day 45
  To evaluate the effect of nirmatrelvir/ritonavir compared to placebo/ritonavir on SARS-CoV-2 viral RNA levels in NP swabs in hospitalized participants.
Incidence of Treatment-Related Adverse Events (TEAEs) | Day 1 through Day 45
  To describe the safety and tolerability of nirmatrelvir/ritonavir relative to placebo/ritonavir for the treatment of severe COVID-19 in hospitalized participants.
Incidence of Adverse Events (AEs) or Serious Adverse Events (SAEs) leading to discontinuations | Day 1 through Day 45
  To describe the safety and tolerability of nirmatrelvir/ritonavir relative to placebo/ritonavir for the treatment of severe COVID-19 in hospitalized participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (2):
  - Bassett Medical Center, Cooperstown, New York
  - Harlem Hospital Center, New York, New York
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment - Sveti Nikolay Chudotvoretz, Lom, Montana
  - Multiprofile Hospital for Active Treatment Sv. Ivan Rilski - Kozloduy EOOD, Kozloduy, Vratsa
  - Multiprofile Hospital for Active Treatment - Haskovo AD, Haskovo
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases - Haskovo EOOD, Haskovo
  - "Specialized Hospital for Active Treatment of Lung Diseases - Pernik" EOOD, Pernik
  - "University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski" EAD, Pleven
  - MHAT - Heart and Brain, Pleven
  - "Multiprofile Hospital for Active Treatment - Medical Complex Sveti Ivan Rilski" EOOD, Plovdiv
  - UMHAT "Prof. Dr. Stoyan Kirkovich"AD, Stara Zagora

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671031